CLINICAL TRIAL: NCT03037359
Title: A Multicenter, Non-interventional, Observational, Prospective Study to Assess Hypotension in Patients With Primary Immunodeficiency Disease Treated With Bivigam™ (Human 10%) or Other Commercial Human 10% Immune Globulin (Intravenous) (IGIV) Products During Infusion and up to 72 Hours Post Infusion
Brief Title: A Study About Low Blood Pressure in Patients With Primary Immunodeficiency Disease Treated With Immune Globulin Products
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ADMA Biologics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 017
Record Dates: First submitted 2017-01-20; First posted 2017-01-31 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Primary Immune Deficiency Disorder
Keywords: PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Immunoglobulin G

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bivigam: Patients with primary immunodeficiency disease treated with Bivigam™
  Interventions: Biological: Bivigam
- Other IGIV: Patients with primary immunodeficiency disease treated with other IGIVs
  Interventions: Biological: Other

INTERVENTIONS:
Biological: Bivigam — Human immune globulin
  Groups: Bivigam
Biological: Other — Human immune globulin
  Groups: Other IGIV

SUMMARY:
This is a safety study to evaluate the risk of low blood pressure in subjects with Primary Immune Deficiency disorder (PID) treated with Bivigam™ or another commercial product under real world conditions. No study medication will be provided to subjects in this study. Study physicians will make all treatment decisions according to their usual practice and will provide prescriptions for his/her subjects, as appropriate. The only addition is the collection and structured documentation of data generated through usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PID diagnosis
* Current subjects requiring treatment with an IGIV

Exclusion Criteria:

* Patients not meeting inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary immunodeficiency disease treated IGIV products.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Hypotension | During infusion and up to 72 hours post infusion.
  The number of events of hypotension in subjects treated with Bivigam or other immune globulin intravenous (IGIV) products.
  Hypotension is defined as a systolic decrease of 30mmHG or a systolic blood pressure less than 90mmHG and clinical symptoms of hypotension including 1 or more of the following: dizziness, light-headedness, fainting (syncope), chest pain, or diaphoresis.

SECONDARY OUTCOMES:
Rate of Hepatic Impairment | Throughout the duration of study participation, up to approximately 140 days.
  The number of events of hepatic impairment in subjects treated with Bivigam or other immune globulin intravenous products. The criterion for defining hepatic impairment is transaminases three times the upper limit of normal evaluated based upon medical history, treatment history and the presence of co-morbid conditions.
Rate of Renal Impairment | Throughout the duration of study participation, up to approximately 140 days.
  The number of events of renal impairment in subjects treated with Bivigam or other immune globulin intravenous. The criterion for defining hepatic impairment is creatinine values greater than three times the upper limit of normal evaluated based upon medical history, treatment history and the presence of co-morbid conditions.
Rates of Other Adverse Events | Throughout the duration of study participation, up to approximately 140 days.
  The rates of other adverse events in patients treated with Bivigam™ or other immune globulin intravenous products.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Santa Barbara Specialty Pharmacy, Carpinteria, California
  - Allergy and Asthma of the Bay Area, Walnut Creek, California
  - Immunoe Research Centers, Centennial, Colorado
  - Central Georgia Infectious Disease Consultants, Macon, Georgia
  - Midwest Allergy and Sinus, Normal, Illinois
  - Kanarek Adult & Pediatric Allergy & Immunology, Overland Park, Kansas
  - Infectious Disease Consultants, Wichita, Kansas
  - The Center for Allergy, Asthma & Immunology, Syosset, New York
  - Allergy Asthma & Immunology Relief, Charlotte, North Carolina
  - Ohio Clinical Research Associates, Mayfield Heights, Ohio
  - Oklahoma Institute of Allergy and Asthma Clinical Research, Oklahoma City, Oklahoma
  - Austin Infectious Disease Consultants, Austin, Texas
  - Discovery Clinical Trials, Dallas, Texas
  - Allergy Partners of North Texas, Dallas, Texas
  - Allergy Immunology and Respiratory Care, Dallas, Texas
  - University of Texas Southwestern Medical Center, Irving, Texas
  - Lysosomal Rare Disorders Research & Treatment Center, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No